CLINICAL TRIAL: NCT01816412
Title: A Prospective, Multicenter, Single Blind, Randomized, Controlled Japanese Population Trial Comparing MD02-LDCB Versus Standard Balloon Angioplasty for Treatment of Femoropopliteal Arteries
Brief Title: LEVANT Japan Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Medicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD02-LDCB
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Femoral Arterial Stenosis; Stenosis of Popliteal Arteries; Femoral Artery Occlusion; Occlusion of Popliteal Arteries
Keywords: Arms; Experimental; Drug Coated Angioplasty Balloon; Active Comparator; Standard angioplasty balloon
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDCB (Experimental): Paclitaxel Coated Balloon
  Interventions: Device: MD02-LDCB Paclitaxel coated balloon catheter
- PTA (Active Comparator): Standard Uncoated Balloon Angioplasty Catheter PTA Catheter
  Interventions: Procedure: Standard Uncoated Balloon Angioplasty Catheter

INTERVENTIONS:
Device: MD02-LDCB Paclitaxel coated balloon catheter
  Arms: LDCB
Procedure: Standard Uncoated Balloon Angioplasty Catheter
  Other Names: PTA Catheter
  Arms: PTA

SUMMARY:
To demonstrate the safety and efficacy of MD02-LDCB for treatment of stenosis or occlusion of the femoral and popliteal arteries in the Japanese population.

DETAILED DESCRIPTION:
The study will enroll patients presenting with claudication or ischemic rest pain and an angiographically significant lesion in the superficial femoral or popliteal artery and a patent outflow artery to the foot. After successful protocol-defined pre-dilatation, subjects that are determined not to require stenting based on defined angiographic criteria are randomized 2:1 to treatment with either MD02-LDCB (test arm) or standard PTA catheter (control arm) using similar techniques. Subjects that do not meet post-predilatation lesion criteria are excluded (and treated per standard practice) and followed for safety for 30 days. Randomized subjects will have ultrasound follow-up through 2 years and are consented for up to 2 years clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ≥20 years of age;
* Rutherford Clinical Category 2-4;
* Length ≤15 cm;
* ≥70% stenosis
* Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the TP trunk;
* A patent inflow artery as confirmed by angiography
* At least one patent native outflow artery to the ankle

Exclusion Criteria:

* Life expectancy of < 2 years;
* History of hemorrhagic stroke within 3 months;
* Previous or planned surgical or interventional procedure within 2 weeks before or within 30 days after the index procedure;
* History of MI, thrombolysis or angina within 2 weeks of enrollment;
* Renal failure or chronic kidney disease
* Severe calcification that renders the lesion un-dilatable

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Composite of freedom from all-cause peri-operative (≤30 day) death and freedom at 6 months from the following: index limb amputation (above or below the ankle), index limb re-intervention, and index-limb-related death. | 6 months
  Primary Patency

SECONDARY OUTCOMES:
Safety | 1, 3, 6, 12 and 24 months
  Composite of freedom from all-cause peri-operative (≤30 day) death and freedom at 6 months from the following: index limb amputation (above or below the ankle), index limb re-intervention, and index-limb-related death.
Efficacy | 1, 3, 6, 12 and 24 months
  Primary Patency of the target lesion at 6 months. Primary Patency is defined as the absence of target lesion restenosis (defined by DUS peak systolic velocity ratio (PSVR) ≥2.5) and freedom from target lesion revascularization (TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyoshi Yokoi, Principal Investigator — Kokura Memorial Hospital Cardiovascular Internal Medicine; Osamu lida, Principal Investigator — Kansai Rosai Hospital Cardiovascular Internal Medicine
Locations (1):
- Kansai Rosai Hospital., Amagasaki-shi, Hyōgo, Japan

REFERENCES:
- [Derived] Ouriel K, Adelman MA, Rosenfield K, Scheinert D, Brodmann M, Pena C, Geraghty P, Lee A, White R, Clair DG. Safety of Paclitaxel-Coated Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2515-2524. doi: 10.1016/j.jcin.2019.08.025. Epub 2019 Sep 28. PMID 31575518